CLINICAL TRIAL: NCT04086810
Title: An Open-Label Study of Diazoxide Choline Controlled-Release Tablet in Patients With Prader-Willi Syndrome
Brief Title: An Open-Label Study of DCCR Tablet in Patients With PWS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study was never initiated; rather the duration of open-label study C602 (NCT03714373) was extended.
Sponsor: Soleno Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C603
Record Dates: First submitted 2019-09-10; First posted 2019-09-12 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2019-09

CONDITIONS: Prader-Willi Syndrome
Keywords: PWS; Prader-Willi Syndrome
MeSH Terms: conditions — Prader-Willi Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DCCR (Experimental): 25 - 450 mg DCCR
  Interventions: Drug: DCCR

INTERVENTIONS:
Drug: DCCR — Once daily oral administration

SUMMARY:
The primary objective of this study is to monitor the long-term safety of DCCR in PWS patients.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of clinical study C602, Visit 15
* Provide voluntary, written informed consent (parent(s) / legal guardian(s) of subject); provide voluntary, written assent (subject, as appropriate)
* Primary caregiver must be able to communicate with Investigator and study site personnel as well as read and complete the study-required questionnaires.

Exclusion Criteria:

* Positive urine pregnancy test (in females of childbearing potential)
* Females who are pregnant or breastfeeding, and/or plan to become pregnant or to breast-feed during or within 90 days after study participation
* Any new disease, condition, or circumstance, which may significantly impact subject safety

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (Safety) | Baseline to Week 106
  Assess the safety of DCCR by evaluating the incidence and severity of adverse events reported.